CLINICAL TRIAL: NCT02804074
Title: MASked-unconTrolled hypERtension Management Based on Office BP or on Out-of-office (Ambulatory) BP Measurement (MASTER Study)
Brief Title: MASked-unconTrolled hypERtension Management Based on Office BP or on Out-of-office (Ambulatory) BP Measurement
Acronym: MASTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: European Society of Hypertension (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09A503
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Masked Hypertension
MeSH Terms: conditions — Masked Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Management strategy of blood pressure based on office BP as a guide to treatment
  Interventions: Other: Optimization of antihypertensive treatment based on office BP
- Group 2 (Experimental): Management strategy of blood pressure based on 24-hour ABPM as a guide to treatment
  Interventions: Other: Optimization of antihypertensive treatment based on 24-hour ABPM

INTERVENTIONS:
Other: Optimization of antihypertensive treatment based on office BP — Optimization of antihypertensive treatment based on office BP
  Arms: Group 1
Other: Optimization of antihypertensive treatment based on 24-hour ABPM — Optimization of antihypertensive treatment based on 24-hour ABPM
  Arms: Group 2

SUMMARY:
MASTER study is a 4-year prospective, randomized, open-label, blinded-endpoint study (PROBE) comparing 2 management strategies 1) office BP as a guide to treatment, or 2) 24-hour ABP as a guide to treatment. Study objectives are to investigate whether a management strategy based on out-of-office BP (Ambulatory BP monitoring) versus a management strategy based on office BP measurements is associated with differences in outcome, including cardiovascular and renal intermediate end points at one year; cardiovascular events at 4 years and changes in a number of blood pressure-related variables throughout the study. Patients will be followed-up during the first year focusing on changes in left ventricular mass index (LVMI, co-primary endpoint) and Urinary albumin excretion (UAE, albumin/creatinine ratio, co-primary end-point), and during the whole 48 month period for both changes in LVMI and UAE and events including all-cause mortality, CV morbidity and mortality, cerebral morbidity and mortality.A total of 1240 subjects will be recruited by 30 centers, taking into account a dropout rate of 15% (620 subjects per randomization arm).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age 35-80 years
* Masked uncontrolled (in treatment) hypertension: office BP <140/90 mmHg, and one or more of the following situations:

  * Ambulatory daytime BP >135/85 mmHg
  * Ambulatory night-time ABP > 120/70 mmHg
  * Ambulatory 24h ABP >130/80 mmHg
* eGFR ≥45 mL/min/1.73 m2 (CKD-EPI creatinine equation 2009)

Exclusion Criteria:

* eGFR <45 mL/min/1.73 m2 (CKD-EPI creatinine equation 2009), and in particular severe chronic renal failure defined as serum creatinine > 250 umol/l;
* Patients in unstable clinical conditions;
* Known secondary hypertension;
* Orthostatic hypotension (SBP fall > 20 mmHg on standing);
* Dementia (clinical diagnosis);
* Hepatic disease as determined by either AST or ALT values > 2 times the upper limit of normal
* History of gastrointestinal surgery or disorders which could interfere with drug absorption
* Known allergy or contraindications to one of the drugs to be administered in the study
* History of malignancy including leukaemia and lymphoma (but not basal cell skin cancer) within the last 5 years
* History of clinically significant autoimmune disorders such as systemic lupus erythematosus.
* History of drug or alcohol abuse within the last 5 years
* History of non-compliance to medical regimens and/or patients who are considered potentially unreliable
* Inability or unwillingness to give free informed consent
* Pregnancy or planned pregnancy during study period.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
changes in LVMI (co-primary endpoint) | 12 months
UAE (albumin/creatinine ratio, co-primary end-point) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Parati, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (2):
- Istituto Auxologico Italiano, Milan, Italy
- Fundacion Venezolana de Hipertension Arterial/Instituto de Enfermedades Cardiovasculares de LUZ, Maracaibo, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Parati G, Agabiti-Rosei E, Bakris GL, Bilo G, Branzi G, Cecchi F, Chrostowska M, De la Sierra A, Domenech M, Dorobantu M, Faria T, Huo Y, Jelakovic B, Kahan T, Konradi A, Laurent S, Li N, Madan K, Mancia G, McManus RJ, Modesti PA, Ochoa JE, Octavio JA, Omboni S, Palatini P, Park JB, Pellegrini D, Perl S, Podoleanu C, Pucci G, Redon J, Renna N, Rhee MY, Rodilla Sala E, Sanchez R, Schmieder R, Soranna D, Stergiou G, Stojanovic M, Tsioufis K, Valsecchi MG, Veglio F, Waisman GD, Wang JG, Wijnmaalen P, Zambon A, Zanchetti A, Zhang Y. MASked-unconTrolled hypERtension management based on office BP or on ambulatory blood pressure measurement (MASTER) Study: a randomised controlled trial protocol. BMJ Open. 2018 Dec 19;8(12):e021038. doi: 10.1136/bmjopen-2017-021038. PMID 30573476